CLINICAL TRIAL: NCT06527950
Title: Analysis of the Anatomical Aspects of the Anterior Mandibular Region for Immediate Implant Placement: An Observational Cone Beam Computed Tomography Study
Brief Title: Anterior Mandibular Region for Immediate Implant Placement
Status: Active, not recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzy Nabil Naiem, Periodontist, Cairo University
Other Study IDs: L123
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — observational study , no intervention

SUMMARY:
Immediate implant placement has been proven to be a successful treatment modality, it is however considered a technique sensitive procedure, which mandates careful planning on basis of the recommended guidelines and thorough site assessment. The anatomical characteristics play a major role in the treatment planning, to determine that enough alveolar bone housing is available to accommodate the implant in the correct prosthetic-driven position and to avoid complications that may be caused by injury of the adjacent anatomical structures. There is scarcity in the literature regarding data on the anatomical features of the mandibular anterior zone in relevance to immediate implant planning. Analysis of the anatomical landmarks of the mandibular anterior region to determine the thickness of the labial and lingual alveolar bony plates, in addition to the bony socket configuration along with the labio-lingual socket dimension and relate them to immediate implant treatment planning

ELIGIBILITY:
Inclusion Criteria:

* CBCTs of teeth including the mandibular anterior zone showing central and lateral incisors and canines.

Exclusion Criteria:

* Radiographs of patients with malaligned teeth or with current or previous orthodontic treatment.
* Radiographs of patients with extensive bone loss due to infection or neoplasm in the area of interest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CBCTs of teeth including the mandibular anterior zone showing central and lateral incisors and canines. The area of interest should include the complete view of roots, alveolar and basal bone related to the centrals, laterals and canines
Sampling Method: Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Labial bone thickness | 1 year
  Linear measurements on CBCT measured in mm

SECONDARY OUTCOMES:
Lingual bone thickness | 1 year
  Linear measurements on CBCT measured in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Giza, Great Cairo, Egypt